CLINICAL TRIAL: NCT06420661
Title: School Partnered Collaborative Care (SPACE) for Pediatric Type 1 Diabetes: A Pilot Feasibility Trial
Brief Title: School Partnered Collaborative Care (SPACE) Intervention for Children With Type 1 Diabetes
Acronym: SPACE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Christine March, Assistant Professor of Pediatrics, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY23120069; K23DK135800 (NIH)
Record Dates: First submitted 2024-05-14; First posted 2024-05-20 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Type 1 Diabetes
Keywords: school; collaborative care model; diabetes care and education; health services
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPACE Intervention (Experimental): The intervention consists of four monthly virtual visits between the school nurse, diabetes care and education specialist (DCES), parent, and any other school-related supports identified by the parent (e.g., coaches, counselors, social workers). At the first visit, the parent and child, school nurse, and DCES will discuss and determine a shared treatment plan. This will include a diabetes medical management plan and shared treatment goals for the child. At each virtual visit, the DCES and school nurse will co-lead the group through review of the shared treatment plan, a review of glucose records and insulin dosing for diabetes management, provide counseling/education, and identify any needed internal (academic) or external (health-related) supports or referrals. Families will be encouraged to set new treatment goals if any milestones are met.
  Interventions: Behavioral: SPACE for T1D
- Control (Active Comparator): In addition to usual care (clinical and in school), parents of children enrolled in the control group will receive four monthly phone calls from the DCES to review diabetes management, mirroring the timing of the virtual visits of the intervention group. This study will employ a wait list control.
  Interventions: Behavioral: Enhanced usual care

INTERVENTIONS:
Behavioral: SPACE for T1D — school-partnered collaborative care model
  Arms: SPACE Intervention
Behavioral: Enhanced usual care — routine diabetes care with optional monthly insulin dose adjustment
  Arms: Control

SUMMARY:
This is a pilot trial of a school-partnered collaborative care (SPACE) model for pediatric type 1 diabetes. The trial will investigate the feasibility and acceptability of SPACE for children with type 1 diabetes in the school setting. SPACE is adapted from a collaborative care model used to treat depression and other mental health care conditions in adolescents and adults.

DETAILED DESCRIPTION:
This pilot cluster randomized controlled trial will examine the feasibility of a school-partnered collaborative care (SPACE) model for children with type 1 diabetes (SPACE for T1D). School districts will be randomized to the intervention or control arm in a 2:1 allocation ratio. School districts randomized to the control arm in Year 1 of the study will be invited to participate in SPACE in Year 2. All children with type 1 diabetes meeting inclusion criteria in each school district will be approached to participate through their school nurse.

All research activities will be conducted using a virtual video-conferencing platform. The intervention arm will consist of four monthly virtual meetings between the child, school nurse, diabetes care and education specialist (DCES), and any other identified school-related support people. The purpose of these meetings will be to determine a shared treatment plan, make treatment recommendations, and determine progress towards meeting the child's goals. The control arm will receive usual care in the school and the clinical setting as well as monthly phone calls from the DCES to the parent to offer review of blood glucoses. No additional contact with the school will be offered.

Participants and their parents will be asked to complete surveys regarding their overall health and well-being and provide us access to their glucometer/continuous glucose monitor data. Additional information will be collected from the electronic health record (hemoglobin A1c, care utilization, referrals). At the end of study, surveys for the parent and school nurse will assess feasibility and other implementation outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 diabetes for at least 6 months
* Attend school in one of the partnered school districts
* Receive daily oversight from the school nurse for their diabetes
* Managed by the Children's Hospital of Pittsburgh Diabetes center
* Able to participate in English

Exclusion Criteria:

* Child has developmental delay or neuropsychiatric disorder which would preclude their participation in their diabetes care and/or completion of study questionnaires
* Child is completely independent in diabetes care in school

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-08-21 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Intervention Measure (FIM) | Month 4
  The primary outcome is feasibility, defined as the extent to which the intervention can be successfully carried out in the school setting. Feasibility will be measured by the FIM, a 4-item scale with an ordinal scoring system from strongly disagree to strongly agree. The scale scores can range from 1-5 with higher scores indicating higher feasibility. The FIM will be completed by the participating child's parent and school nurse. The school nurses will be asked to complete the measure for each iteration of SPACE, which will mean that the same nurse may complete the measure multiple times. Nurses will need to complete the measure within 14 days of the end of that iteration of SPACE, allowing us to descriptively assess change in an individual school nurse's response over time. The intervention will be deemed "feasible" if the mean overall score is >4/5 (80%).

SECONDARY OUTCOMES:
Acceptability of Intervention Measure (AIM) | Month 4
  Acceptability is defined as the perception that the intervention is agreeable or satisfactory. Acceptability will be measured with AIM, a 4-item scale with an ordinal scoring system from strongly disagree to strongly agree. The scale scores can range from 1-5 with higher scores indicating higher acceptability. The AIM will be completed by the participating child's parent and school nurse. The school nurses will be asked to complete the measure for each iteration of SPACE, which will mean that the same nurse may complete the measure multiple times. Nurses will need to complete the measure within 14 days of the end of that iteration of SPACE, allowing us to descriptively assess change in an individual school nurse's response over time. The intervention will be deemed "acceptable" if the mean overall score is >4/5 (80%).
Intervention Appropriateness Measure (IAM) | Month 4
  Appropriateness is defined as the perceived fit or relevance of the intervention to the school setting. Appropriateness will be measured with the IAM, a 4-item scale with an ordinal scoring system from strongly disagree to strongly agree. The scale scores can range from 1-5 with higher scores indicating higher appropriateness. The IAM will be completed by the participating child's parent and school nurse. The school nurses will be asked to complete the measure for each iteration of SPACE, which will mean that the same nurse may complete the measure multiple times. Nurses will need to complete the measure within 14 days of the end of that iteration of SPACE, allowing us to descriptively assess change in an individual school nurse's response over time. The intervention will be deemed "appropriate" if the mean overall score is >4/5 (80%).
Intervention Usability Scale (IUS) | Month 4
  Usability is defined as the degree to which the intervention is able to be used. Usability will be measured by the IUS, a 10-item scale with an ordinal scoring system from strongly disagree to strongly agree. The scale scores can range from 1-5 with higher scores indicating higher usability. The IUS will be completed by the participating child's parent and school nurse. The school nurses will be asked to complete the measure for each iteration of SPACE, which will mean that the same nurse may complete the measure multiple times. Nurses will need to complete the measure within 14 days of the end of that iteration of SPACE, allowing us to descriptively assess change in an individual school nurse's response over time. The intervention will be deemed "usable" if the mean overall score is >4/5 (80%).

CONTACTS AND LOCATIONS:
Overall Officials: Christine A March, MD, Principal Investigator — Univeristy of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No